CLINICAL TRIAL: NCT04981743
Title: Evaluation of The Efficacy of Nigella Sativa Versus VitaminD3 as Supplement Therapy in Management of Coronavirus Disease 2019 (COVID-19)
Brief Title: The Efficacy of Nigella Sativa Versus VitaminD3 as Supplement Therapy in Coronavirus Disease 2019 (COVID-19)
Acronym: COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: supplement therapy in COVID-19
Record Dates: First submitted 2021-07-09; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Controlled Parallel Open label Randomized Clinical Trial .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (No Intervention): Twenty five patients will be administered only the standard treatment regimen according to Ministry Of Health, and Population management protocol for COVID-19 patients (November 2020).
- group 2 (Active Comparator): Twenty five patients will be administered a single dose (900mg) of Nigella Sativa capsule twice daily plus standard therapy
  Interventions: Dietary Supplement: Nigella Sativa capsule twice daily
- group 3 (Active Comparator): Twenty five patients will be administered a single dose (2000 IU) of vitamin D3 tablet once daily plus standard therapy
  Interventions: Dietary Supplement: Nigella Sativa capsule twice daily
- group 4 (Active Comparator): Twenty five patients will be administered a single dose (900 mg) of Nigella Sativa capsule twice daily, and single dose of vitamin D3 tablet (2000 IU) once daily plus standard therapy.
  Interventions: Dietary Supplement: Nigella Sativa capsule twice daily

INTERVENTIONS:
Dietary Supplement: Nigella Sativa capsule twice daily — investigate the safety and efficacy of Nigella Sativa versus Vitamin D3 versus Nigella Sativa / vitamin D3 combination as supplement for management of COVID-19 .
  Other Names: single dose of vitamin D3 tablet (2000 IU) once daily
  Arms: group 2; group 3; group 4

SUMMARY:
The aim this study is to investigate the safety and efficacy of Nigella Sativa versus Vitamin D3 versus Nigella Sativa / vitamin D3 combination as supplement for management of COVID-19 .

DETAILED DESCRIPTION:
Corona-virus disease-19 (COVID-19) is caused by the severe acute respiratory syndrome coronavirus 2, and this virus was first originated from Wuhan city of Hubei province of China spreading around the globe. The prominent symptoms of COVID-19 include fever, cough, dyspnea, and other symptoms noted in patients affected by COVID-19 that includes; chills, repeated shaking with chills, muscle pain, headache, sore throat, and new loss of taste or smell. In addition, the emergency warning signs of COVID-19 include difficulty breathing or shortness of breath, persistent pain or pressure in the chest, new confusion or inability to arouse and bluish lips or face and the patients experiencing any of these signs should get immediate medical attention.

Herbal medicines are used by many people to try to improve their health upon the believe that "natural products" are always safe, and good for immunity based on the traditional knowledge .There is a potential of Nigella Sativa to treat the patients with COVID-19.

Nigella Sativa (NS), a widely used medicinal plant of the family Ranunculaceae ; commonly known as Black Cumin, has been shown to exert antiviral effects against a variety of viruses such as Mouse Cytomegalovirus and Hepatitis C Virus (HCV) . The components' antimicrobial properties against various microbes as well as their anti-inflammatory and immuno-modulatory effects have also been established .

The immune system defends the body from foreign, invading organisms, promoting protective immunity, while maintaining tolerance to self. The implications of vitamin deficiency on the immune system have become clearer in recent years, and in the context of vitamin D deficiency, the increased susceptibility to infection observed, especially in a genetically susceptible host to autoimmunity.

The classical actions of vitamin D are to promote calcium homeostasis, and to promote bone health. In humans, vitamin D is obtained from the diet, or synthesized in the skin as vitamin D is cutaneously produced after exposure to UV light, its synthesis is influenced by latitude, season, use of sun-block and skin pigmentation. Melanin absorbs UV radiation inhibiting the synthesis of vitamin D from 7-dihydrocholesterol. This initial vitamin D compound is inactive form; hydroxylation in the liver to form the active 25 hydroxy vitamin D3 (25 D). Vitamin D is the most reliable measurement of an individual's vitamin D status. It is converted in the kidney to the active compound 1,25 dihydroxy vitamin D (1,25 D) or calcidiol by 1-α-hydroxylase (CYP27B1), an enzyme which is stimulated by parathormone.

A principal defense against uncontrolled inflammation, and against viral infection in general, is provided by T regulatory lymphocytes (Tregs). Treg levels have been reported to be low in many COVID-19 patients, and can be increased by vitamin D supplementation. Low vitamin D levels have been associated with an increase in inflammatory cytokines, and a significantly increased risk of pneumonia, and viral upper respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild-moderate COVID-19 according to the classification (Table 1)
2. Adult (18 - 65 years old).
3. Polymerase chain reaction (PCR)-confirmed infection with Severe Acute Respiratory Syndrome Coronavirus-2.

Exclusion Criteria:

1. Patients with severe illness requiring admission to intensive care unit.
2. Asymptomatic patients.
3. Severe chronic kidney disease (i.e. estimated glomerular filtration rate < 30 mL/min) or end stage renal disease requiring dialysis
4. Severe chronic liver disease (Alanine transaminase or Aspartate transaminase > 5 times the upper limit of normal).
5. contraindications to any of the interventional drugs.
6. Pregnancy or breast feeding.
7. Allergy to any of the interventional.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-21 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The safety and efficacy of Nigella Sativa and Vitamin D3 as a supplement for management of COVID-19 will be evaluated and recorded. | baseline and 14 days
  The patient will be examined by the physician and the rate of occurrence of any of the following signs and symptoms on the participants will be reported:
  * Fever -Runny nose - Red swollen eyes
  * Fatigue - Shortening in breath - Skin rash
  * Cough - Body aches
  * Sore throat - Diarrhea, and/or Vomiting
  * Headache - Loss of taste and/or Smell
Assessment of patient health status before and after treatment intervention for a period of 14 days will be done | baseline and 14 days
  All patients will be evaluated during the study period (14 days) by undergoing PCR test after two days from absence of any clinical presentation, Then if the PCR is negative, the patient will be discharged from the hospital and complete his medication course at home.
  * If the result is positive then the patient will undergo another PCR testing on day 14 with no further follow up .

SECONDARY OUTCOMES:
The recovery rate of patients, Intensive care unit admission rate of patients and the Length of hospital stay of the patients will be recorded | 14 days
  Length of hospital stay and number of patients need ICU admission due to deterioration of cases and progression of disease.
The following laboratory testing will be performed at least twice during the study period: | 14 days
  * C-Reactive Protein in mg/L.
  * Arterial Blood Gases[carbon dioxide partial pressure, oxygen partial pressure] in mm Hg.
  * Kidney function [serum creatinine, blood urea nitrogen ] in mg/dL.
  * liver function [ Alanine aminotransferase, Aspartate aminotransferase] in IU/L .
  * Erythrocyte sedimentation rate in mm/hr.
  * Complete blood picture.
  * Serum Ferritin in ug/L
  * international normalized ratio, prothrombin time, partial thromboplastin time in seconds
  * Polymerase chain reaction (PCR).
  * Computed tomography (CT) chest .
  Length of hospital stay and number of patients need ICU admission due to deterioration of cases and progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A. Sabri, professor, Study Chair — Department of Clinical Pharmacy
Locations (1):
- Respiratory System specialized hospital at Kobry Elobba Military Medical hospitals., Cairo, Egypt

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Horowitz RI, Freeman PR, Bruzzese J. Efficacy of glutathione therapy in relieving dyspnea associated with COVID-19 pneumonia: A report of 2 cases. Respir Med Case Rep. 2020 Apr 21;30:101063. doi: 10.1016/j.rmcr.2020.101063. eCollection 2020. PMID 32322478
- [Background] Montero-Odasso M, Goens SD, Kamkar N, Lam R, Madden K, Molnar F, Speechley M, Stranges S. Canadian Geriatrics Society COVID-19 Recommendations for Older Adults. What Do Older Adults Need To Know? Can Geriatr J. 2020 Mar 1;23(1):149-151. doi: 10.5770/cgj.23.443. eCollection 2020 Mar. No abstract available. PMID 32269670
- [Derived] Said SA, Abdulbaset A, El-Kholy AA, Besckales O, Sabri NA. The effect of Ni gella sativa and vitamin D3 supplementation on the clinical outcome in COVID-19 patients: A randomized controlled clinical trial. Front Pharmacol. 2022 Nov 8;13:1011522. doi: 10.3389/fphar.2022.1011522. eCollection 2022. PMID 36425571